CLINICAL TRIAL: NCT05402696
Title: The St. Paul's Hospital Advanced Endoscopic Resection Centre Cohort for Colorectal Neoplasia (SPARC-C): A Prospective Observational Study
Brief Title: St. Paul's Advanced Resection Center Cohort for Colorectal Neoplasia (SPARC-C)
Acronym: SPARC-C
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Neal Shahidi, Assistant Professor of Medicine, University of British Columbia
Other Study IDs: H22-00037
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Colon Adenoma; Colon Polyp; Colon Lesion
Keywords: Colorectal neoplasia; Advanced endoscopy; Endoscopic resection
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Large non-pedunculated colorectal polyp (LNPCP): Patients referred to St. Paul's Hospital for endoscopic management of a large (≥20mm) non-pedunculated colorectal polyp (LNPCP).
  Interventions: Procedure: Endoscopic tissue resection

INTERVENTIONS:
Procedure: Endoscopic tissue resection — Endoscopic resection techniques for removal of large polyps
  Other Names: Endoscopic mucosal resection; Endoscopic submucosal dissection; Colonoscopic polypectomy

SUMMARY:
The SPARC-C study is a prospective, single-centre observational study of patients referred for the management of large (≥ 20mm) non-pedunculated colorectal polyps (LNPCPs). Patients are managed consistent with current standards of care. Prospectively collected data includes: patient clinicodemographic details, lesion details, procedural details, and clinical outcomes.

DETAILED DESCRIPTION:
Endoscopic resection techniques, including endoscopic mucosal resection (EMR), endoscopic submucosal dissection (ESD), and cold snare resection (CSR), have become the primary treatment strategy for the vast majority of large non-pedunculated colorectal polyps (LNPCPs). This is because of the efficacy, safety, and cost-effectiveness of endoscopic techniques compared to surgery. Site-specific technical modifications and the development of auxiliary techniques/strategies have mitigated the risk of technical failure, clinically significant post-resection bleeding (CSPEB), significant deep mural injury (S-DMI)/perforation, and recurrence. However, questions still remain about the application and selection of these techniques.

This is a single-centre cohort study of consecutive patients referred for the management of LNPCPs to one of two interventional endoscopists with a tertiary referral practice in minimally invasive endoscopic resection techniques. It is based at St. Paul's Hospital and its affiliated sites, with the aim of enrolling 3500 participants over 10 years.

This cohort serves as a platform to continue refining the management of LNPCPs. We will evaluate LNPCP management outcomes, including technical success, clinical success, clinically significant intra-procedural bleeding (CSIPB), S-DMI, CSPEB, delayed perforation, recurrence, and referral to surgery. Findings will also help to further refine mitigating strategies for intra-procedural and post-procedural adverse outcomes (CSPIB, S-DMI, CSPEB, delayed perforation, recurrence, and referral to surgery). Finally, we aim to optimize the application of minimally invasive endoscopic resection techniques for the management of LNPCPs, including the development of artificial intelligence clinical decision support solutions (AI-CDSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age referred for the management of an LNPCP
* Able to provide informed consent.

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age who have been referred to St. Paul's Hospital from 2022 to 2032 for management of a large (≥20mm) non-pedunculated colorectal polyp (LNPCP).
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical Success of Endoscopic Procedure | Intra-procedure
  Complete removal of all visible polypoid tissue during index procedure.
Clinical Success of Endoscopic Procedure | 6 months
  Technical success and the avoidance of surgery for large non-pedunculated colorectal polyps (LNPCPs) referred for endoscopic resection, assessed at first surveillance colonoscopy. LNPCPs with features consistent with invasive disease and directly referred for surgery are excluded.

SECONDARY OUTCOMES:
Peri-Procedural Adverse Outcomes | 6 months
  Frequency and management of peri-procedural adverse outcomes including clinically significant intra-procedural bleeding, significant deep mural injury, clinically significant post-resection bleeding, delayed perforation, recurrence, and referral to surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Mount Saint Joseph Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Pacific Gastroenterology Associates, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No